CLINICAL TRIAL: NCT06863051
Title: Clinical and Radiographic Evaluation of Xenograft With Albumin Platelet-Rich Fibrin or Leucocyte- Platelet-Rich Fibrin on Immediate Implant Placement in Mandibular Molar Extraction Sites: Randomized Clinical Trial.
Brief Title: Effect of Albumin Platelet-Rich Fibrin or Leucocyte- Platelet-Rich Fibrin on Immediate Implant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mostafa Fayed, Demonstrator of Periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-531
Record Dates: First submitted 2025-02-27; First posted 2025-03-07 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Immediate Implant Placement
Keywords: Implant; PRF; Albumin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin-PRF group (Experimental): Immediate Implant Placement in lower molar region, Grafted with Xenograft and Albumin PRF Gel
  Interventions: Procedure: Immediate Implant Placement and Alb-PRF
- L-PRF group (Experimental): Immediate Implant Placement in lower molar region, Grafted with Xenograft and L-PRF ( L-PRF Block )
  Interventions: Procedure: Immediate Implant Placement and L-PRF

INTERVENTIONS:
Procedure: Immediate Implant Placement and Alb-PRF — Immediate Implant Placement in lower molar region, Grafted with Xenograft and Albumin PRF Gel
  Arms: Albumin-PRF group
Procedure: Immediate Implant Placement and L-PRF — Immediate Implant Placement in lower molar region, Grafted with Xenograft and L-PRF
  Arms: L-PRF group

SUMMARY:
The objective of this study will be to compare between Immediate Implant grafted with xenograft and Alb-PRF gel versus xenograft with L-PRF.

DETAILED DESCRIPTION:
The objective of this study will be to compare between xenograft with Alb-PRF gel and xenograft with L-PRF ( L-PRF Block ) in the aspects of :

* Peri-implant vertical defect depth.
* Crestal bone level.
* Bucco-lingual bone width.
* Keratinized tissue width

ELIGIBILITY:
1. Inclusion criteria

   * The presence of non-restorable mandibular molar.
   * Patient 18-45 years old
   * Intact buccal and lingual walls
   * Good oral hygiene.
   * Prescence of sufficient restorative space.
   * Jumping gap more than 2 mm.
2. Exclusion criteria

   * Proximity of anatomical structures
   * Acute localized infection (suppuration at the surgical field)
   * Patients on chemotherapy or radiotherapy.
   * Patients who have systemic disorders (diseases) {diabetes mellitus, autoimmune disease, …etc},
   * Pregnant patients.
   * Smoking and Alcohols.
   * Presence of periapical pathology affecting the neighboring teeth.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Vertical peri-implant bone level | Immediate Post-Operative and 6 months after surgery
  the distance between implant platform to the most coronal bone-implant contact
Keratinized tissue Width | Immediate Post-Operative and 6 months after surgery
  Width of Keratinized tissue before and after surgery
Crestal bone level | Immediate Post-Operative and 6 months after surgery
  distance between implant platform and bone crest

SECONDARY OUTCOMES:
Implant Stability | Immediate Post-Operative and 6 months after surgery
  by Smart peg
Bucco-lingual bone width | Immediate Post-Operative and 6 months after surgery
  it's measured with a line coinciding with implant platform

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Faculty of Dentistry, Kafr ash Shaykh, Kafrelsheikh, Egypt